CLINICAL TRIAL: NCT04854161
Title: Online Training of Empathic Attunement to Affect: the Impact of Compassion
Brief Title: Online Training of Empathic Attunement to Affect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UPC-21-02-Compassi-ON
Record Dates: First submitted 2021-03-04; First posted 2021-04-22 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-05

CONDITIONS: Empathy
Keywords: Clinical Trial Protocols

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compassion and Empathic Attunement to Affect (Experimental): Empathic Attunement to Affect is based on Emotion-Focused Therapy. Compassion training program is based on Compassion Cultivation Training, CCT
  Interventions: Behavioral: Empathic Attunement to Affect Training; Behavioral: Compassion Training
- Focusing and Empathic Attunement to Affect (Active Comparator): Empathic Attunement to Affect is based on Emotion-Focused Therapy. Focusing training program is based on Focusing-Oriented Therapy
  Interventions: Behavioral: Empathic Attunement to Affect Training; Behavioral: Focusing Oriented Therapy Training

INTERVENTIONS:
Behavioral: Empathic Attunement to Affect Training — Empathic Attunement to Affect:
  Empathy and neuroscience Therapeutic Presence
  Opening receptivity channels Empathic reflections and landscapes (external, meaning and feeling)
  Types of emotions: Primary (adaptive, maladaptive), Secondary. Emotion Scheme Types of experiential responses: conjectures, exploration.
  Working with Core emotions Types of experiential responses: Evocation and Empathic affirmation,
  Empathy and Emotion Productivity Types of experiential responses: Empathic formulation, process suggestion Difficult situations: working on assertive anger and self-soothing Types of experiential responses: Facilitative Congruence
Behavioral: Compassion Training — Compassion Training Introduction to Mindfulness Compassion toward a significant other Compassion toward a generic other Self-compassion Tonglen Compassion toward a difficult other
  Arms: Compassion and Empathic Attunement to Affect
Behavioral: Focusing Oriented Therapy Training — Focusing-Oriented Therapy training Introduction to focusing Acceptance and empathy as the main focusing attitudes Fels-sense markers Felt sense, handle and resonance Hakomi Therapy The Safe Place. Focusing with a challenging person
  Arms: Focusing and Empathic Attunement to Affect

SUMMARY:
TThis research wants to observe the effectiveness of an Empathic attunement online training program for psychologists. This training is based on emotion-focused therapy.

The present research has one main objective and two secondary objectives. The main objective of is to explore the impact of compassion training as a facilitator of empathic attunement training. For this reason, an experimental design will be conducted, randomly assigning therapists to two training programs on empathy, one of them accompanied by compassion training and the other accompanied by focusing training.

Secondary objectives:

* To validate in Spanish three empathy measures, the empathic understanding subscale from Barrett-Lennard´s relational inventory, Watson´s Observation of expressed empathy measure and the empathy subscale made from the Sussex-Oxford Compassion for Others Scale.
* To explore patient variables related to empathy perception, especially the role of self-critic.

DETAILED DESCRIPTION:
This research wants to observe the effectiveness of an Empathic attunement online training program for psychologists. This training is based on emotion-focused therapy.

The present research has one main objective and two secondary objectives. The main objective of is to explore the impact of compassion training as a facilitator of empathic attunement training. For this reason, an experimental design will be conducted, randomly assigning therapists to two training programs on empathy, one of them accompanied by compassion training and the other accompanied by focusing training.

Secondary objectives:

* To validate in Spanish three empathy measures, the empathic understanding subscale from Barrett-Lennard´s relational inventory, Watson´s Observation of expressed empathy measure and the empathy subscale made from the Sussex-Oxford Compassion for Others Scale (SOCS-O).
* To explore patient variables related to empathy perception, especially the role of self-critic.

Detailed Description

Objectives and hypothesis

I. The main objective of the present paper: Explore the impact of compassion empathy on an empathic attunement training program.

The following hypothesis will be contrasted:

1. Presumably, the training on empathy/compassion will increase therapeutic presence to a larger extent than the empathy/focusing training. A statistically significant effect of the interaction of time x group on presence scores is expected.
2. Presumably, the training on empathy/ compassion will increase the emotional regulation abilities of the therapists to a larger extent than the empathy/focusing training. A statistically significant effect of the interaction of time x group on the DERS subscales ratings is expected.
3. Presumably, the empathy/compassion training will increase the therapists therapeutic Alliance scoring to a larger extent than the empathy/focusing training. A statistically significant effect of the interaction of time x group on the alliance scoring is expected.
4. Presumably, the empathy/compassion training will reduce empathic distress (Interpersonal Reactivity Index) and the empathic distress (Cognitive and Emotional Empathy Test), it will increase empathic happiness (Cognitive and Emotional Empathy Test) and the empathic worry (Interpersonal Reactivity Index) to a larger extent than the empathy/focusing training. A statistically significant effect of the interaction of time x group on these measures is expected. Specifically on the Interpersonal Reactivity Index and Cognitive and Emotional Empathy Test subscales scores. On the other hand, fantasy (Interpersonal Reactivity Index), empathic perspective (Interpersonal Reactivity Index), perspective adoption (Cognitive and Emotional Empathy Test) and emotional understanding (Cognitive and Emotional Empathy Test), are expected to remain unchanged on both empathy training groups.
5. Mediation hypothesis: Changes of the therapist's empathy (Cognitive and Emotional Empathy Test, Interpersonal Reactivity Index, empathic understanding, expressed empathy) on empathy/compassion compared to empathy/focusing, will be mediated by changes on facets of mindfulness (Five Facet Mindfulness Questionnaire) and self-compassion (Self-Compassion Scale; Sussex-Oxford Compassion Scale).

II. Spanish validation of empathy measures (empathic understanding subscale from Barrett-Lennard´s relational inventory, expressed empathy, and the Sussex-Oxford Compassion Scale.

1. Criterion Validity: Statistically significant correlation between the expressed empathy measure and empathic understanding measures are expected. Significant correlations between self-report measures (Interpersonal Reactivity Index, Cognitive and Emotional Empathy Test) and the measures of expressed empathy and the empathic understanding measures, as well as therapeutic presence, are expected.
2. Evidence for adequate reliability (Cronbach´s alfa and McDonald´s omega) on the empathic understanding measures of the relational inventory, both on the therapists and the patient's version, is expected.
3. Evidence for an adequate interrater reliability on the expressed empathy measures is expected.
4. Incremental validity: The patient's version of empathic understanding explain will show statistically significant associations with the session evaluation (alliance), once controlled the empathic understanding assessed by the therapists and expressed empathy (assessed by external raters). However, the empathic understanding version of the therapist will not explain variance once discounted the effect of the patient's version and expressed empathy.

III. Explore patient variables related to empathy evaluation: the role of patient´s self-critic.

1. Empathy perceived by patients with higher self-critic scoring will be inferior to the empathy perceived by patients with less self-critic scoring.
2. Empathy/compassion training will get higher scores on these patients than the empathy/focusing training.

Recruitment

Phase 1:

To recruit people as patients, students from Comillas University will be asked to participate, coming from Psychology and other degrees. They will be informed about the research goals, as well as their role and personal data protection. If they wish to participate, they will be asked to sign an informed consent to use the data and ask them to facilitate their email so they can be contacted, and self-critic questionnaire will be administered.

In every moment participants will have available the contact information of the main researcher so they can ask any question or doubt. Participants will also be informed that they can revoke their participation and the storage of their data at any moment.

Regarding the therapists, a brochure will be disseminated on social networks with all the information about the research.

Phase 2:

Patients and therapists will receive an email, with all the information about the research development and will be asked to sign the informed consent about the usage of their information, as well as a specific confidentiality document for the therapists about the information they are going to gather from the patients during the online interview.

Participants

1. Therapists in training Based on previous meta-analysis, we predict a mean effect size (g of Hedge=0.51) on the change between previous and subsequent moments to treatment. A power analysis assuming an alfa of 0.05, with a potency of 0.8, reveals that 26 participants are necessary. A total of 30 participants for each condition is aimed in this study.

   To handle the high drop-out rate, usually present in online interventions, 80 therapists will be randomly allocated between two conditions: compassion training and focusing training.

   Exclusion criteria for the therapists group: every student that has taken the "empathic attunement" course will be excluded. Subjects that have received training in either focusing or compassion will also be excluded.

   Inclusion criteria for the therapists group: Psychologists with experience in Psychotherapy (at least one client).
2. Participants interviewed as patients A total of 40 people will be interviewed by the therapists. Exclusion criteria for participants/patients: Participants presenting severe mental illness (schizophrenia, psychotic and personality disorders) will be excluded, those presenting severe addictions or eating disorders will also be excluded. The presence of these diagnoses will be inquired.

Inclusion criteria for participants/patients: voluntary participation, above 18 years-old

• Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing: Two external experts will monitor and audit the research project, and data registry.

Method Once the voluntary therapists are inscribed, they will be randomized on one randomizing session using sample function to generate random numbers on R statistical package.

The therapists in training who participate will receive the measures exposed on table 2.

Therapist self-report measures. Pre and post self-report measures: Cognitive and Emotional Empathy Test, Interpersonal Reactivity Index, Self-Compassion Scale, Five Facet Mindfulness Questionnaire, Sussex-Oxford Compassion Scale Measures after the pre and post interview: Presence and RI, Adherence to program measures

With this group of measures affective, cognitive and behavioral aspects of empathy are encompassed. Participants on the patient's role will receive the measures depicted on Table 3. Two external judges will evaluate the 10 final minutes of the intervention, evaluating the expressed empathy of the therapist.

Table 3. Self- report measures for the participants on the patient role. BAI FSCRS RI-EU therapist empathy (patient version) Therapist presence (patient version) SRS (session evaluation)

Interview method To make the interview, each patient and therapist will receive and appointment by means of an online Teams session, to ensure data confidentiality.

To simulate a psychotherapy session, and activate emotional processes previous to the empathic exploration, the participant will be invited to do a two-chair dialogue to explore his/her self-critic voice and his/her experiencing voice. Lastly, the therapist is asked to explore empathically for 20 minutes.

Data analysis

Mixed linear models will be used to analyze the impact of different types of training on the dependent variables analyzed. The statistical package lme4 will be used (Bates, Mächler, Bolker and Walker, 2015), of R (R Core Team, 2020).

The mediation analysis will be done using SPSS and the process syntax of Hayes (2017).

Working with adherence criterion: Participants that do not attend more than a 25% of the sessions will be eliminated. G * Power 3.1. 9. 6 (Faul, Erdfelder, Lang, and Buchner, 2007) was used for the potency calculations.

ELIGIBILITY:
Inclusion Criteria:

* Psychologists with experience in psychotherapy (at least one client)

Exclusion Criteria:

* Previous empathic attunement training
* Previous Compassion training
* Previous Focusing training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Cognitive and affective empathy test | 5 minutes
  TECA; López-Pérez, Fernández-Pinto and Abad, 2008. Scores range from 33 to 132, with higher values reflecting higher empathy.
Interpersonal reactivity index | 5 minutes
  IRI; Davis, 1980. Scores range from 28 to 140, with higher values reflecting higher empathy.
Empathic Understanding of Relationship Inventory | 3 minutes
  EU; Barrett-Lennard (1986). Scores range from -48 to 48, with higher values reflecting higher empathy
Expressed Empathy Inventory | 20 minutes
  Watson, 1999. Scores range from 0 to 9, with higher values reflecting higher empathy

SECONDARY OUTCOMES:
Self-Compassion Scale | 5 minutes
  SCS; Neff, 2003; Translated and validated into Spanish population by García-Campayo et al., 2014. Scores range from 26 to 130, with higher values reflecting higher compassion.
Five Facet Mindfulness Questionnaire | 5 minutes
  Baer, Smith, Hopkins, Krietemeyer y Toney, 2006), the Spanish version (Cebolla, García-Palacios, Soler, Guillen, Baños and Botella, 2012). Scores range from 39 to 195, with higher values reflecting higher mindfulness trait.
Compassion scales of Sussex-Oxford | 5 minutes
  SOCS; Gu, Baer, Cavanagh, Kuyken, and Strauss, 2020. Scores range from 20 to 100, with higher values reflecting higher compassion.

OTHER OUTCOMES:
Session Rating Scale | 1 minute
  Short therapeutic alliance measure. (Duncan et al., 2003; Gismero and Cagigal, 2020).Scores range from 0 to 10, with higher values reflecting higher working alliance.
Difficulties in emotional regulation | 5 minutes
  DERS; Gratz and Roemer, 2004; Hervás and Jódar, 2008. Scores range from 36 to 180, with higher values reflecting lower emotional regulation.
Therapeutic presence | 3 minutes
  Geller et al., 2010; Martín-Íñigo, 2015. Scores range from 21 to 105, with higher values reflecting higher presence.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Jódar Anchía, Study Director — Universidad Pontificia Comillas; Carlota Martín, Principal Investigator — Universidad Pontificia Comillas
Locations (1):
- Comillas Pontifical University, Madrid, Spain